CLINICAL TRIAL: NCT06162962
Title: Department of Orthopedic Oncology, The First Affiliated Hospital of Sun Yat-sen University
Brief Title: Oncological and Functional Outcomes in Lower Limb Osteosarcoma Pediatric Patient
Status: Completed | Type: Observational
Sponsor: Changye Zou (Other)
Responsible Party: Sponsor-Investigator, Changye Zou, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: Changye Zou
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Osteosarcoma; Pediatric; Lower Limb Injury; Outcome
MeSH Terms: conditions — Osteosarcoma; Leg Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- age groups: The general characteristic of patients and clinical data including age, Enneking stage, surgical methods, type of prosthesis, primary tumor location were recorded.
  Interventions: Other: Retrospective analysis
- surgical methods: The general characteristic of patients and clinical data including age, Enneking stage, surgical methods, type of prosthesis, primary tumor location were recorded.
  Interventions: Other: Retrospective analysis
- type of prosthesis: The general characteristic of patients and clinical data including age, Enneking stage, surgical methods, type of prosthesis, primary tumor location were recorded.
  Interventions: Other: Retrospective analysis
- primary tumor location: The general characteristic of patients and clinical data including age, Enneking stage, surgical methods, type of prosthesis, primary tumor location were recorded.
  Interventions: Other: Retrospective analysis
- Enneking stage: The general characteristic of patients and clinical data including age, Enneking stage, surgical methods, type of prosthesis, primary tumor location were recorded.
  Interventions: Other: Retrospective analysis

INTERVENTIONS:
Other: Retrospective analysis — Retrospective analysis

SUMMARY:
Retrospective analysis of specific characteristics of complications and long-term oncological and function outcomes in lower-limb osteosarcoma pediatric patients.

DETAILED DESCRIPTION:
Clinical and functional outcomes were compared based on age groups, surgical methods, type of prosthesis, and primary tumor location. Patients were divided into the Low-age group (≤10 years old) and the High-age group (>10 years old). Overall Survival rate (OS), Progression-Free Survival rate (PFS), and prosthesis survival rate were assessed using Kaplan-Meier curves, and non-parametric survival analysis (log-rank test) was used for comparison. The incidence of complications, local relapse rate (LRR), metastasis rate, final limb-salvage and amputation rate, and Musculoskeletal Tumor Society (MSTS) score of different independent groups were further evaluated using χ2 test or Fisher's exact test, and t-test was employed to evaluate the measurement data.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed lower limb osteosarcoma patients under the age of 14;
2. Performing tumor resection treatment in our hospital;
3. There is complete clinical registration data available.

Exclusion Criteria:

1. Not undergoing surgical treatment in our hospital;
2. Age older than 14 years old;
3. No available clinical registration data or lost follow-up patients;
4. Non lower limb osteosarcoma patients.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A retrospective analysis of 345 pediatric patients with lower-limb osteosarcoma admitted to our department between 2000 and 2019 was conducted.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Overall Survival rate (OS) | 2000-2019
  Oncological outcomes
Progression-Free Survival rate (PFS) | 2000-2019
  Oncological outcomes
Local recurrence rate(LRR) | 2000-2019
  Oncological outcomes
Metastasis rate | 2000-2019
  Oncological outcomes
Final limb-salvage and amputation rate | 2000-2019
  Oncological outcomes
Prosthesis survival rate | 2000-2019
  Functional outcomes
Musculoskeletal Tumor Society (MSTS) score | 2000-2019
  Functional outcomes
Complications | 2000-2019
  Functional outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Changye Zou, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets are available from the corresponding author (zouchy@mail.sysu.edu.cn) on reasonable request after SCI online.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: SCI online. The datasets are available from the corresponding author on reasonable request.
Access Criteria: The datasets are available from the corresponding author (zouchy@mail.sysu.edu.cn) on reasonable request after SCI online.

REFERENCES:
- [Derived] Xu M, Tu J, Huang Y, Wang B, Zhao Z, Lin T, Huang G, Yin J, Xie X, Shen J, Zou C. Comparison of oncological and functional outcomes in Lower-limb osteosarcoma pediatric patients: a large single-center retrospective cohort study. Int J Surg. 2024 Jul 1;110(7):4208-4220. doi: 10.1097/JS9.0000000000001340. PMID 38471042